CLINICAL TRIAL: NCT04572399
Title: Respiratory Application of a Novel Ultraviolet Light Delivery Device for Patients Infected With COVID-19: A Pilot Study
Brief Title: UVA Light Device to Treat COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Aytu BioPharma, Inc. (Industry)
Responsible Party: Principal Investigator, George Chaux, Medical Director, Lung Transplant Program, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 883
Record Dates: First submitted 2020-09-28; First posted 2020-10-01 (Actual); Results first posted 2022-01-18 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Intubated patients with confirmed SARS-CoV-2 will receive UV light treatment to potentially reduce bacterial and viral burden.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Endotracheal UV Light (Experimental): Mechanically ventilated patients who will receive UV Light therapy
  Interventions: Device: UV Light Treatment

INTERVENTIONS:
Device: UV Light Treatment — UV light therapy administered while patient is mechanically ventilated

SUMMARY:
This pilot study will assess the safety and effectiveness of UV light treatment in hospitalized patients with COVID-19.

DETAILED DESCRIPTION:
This is a single center, open label, pilot study. 5 adult patients, aged over 18, who are confirmed positive with SARS-CoV-2 and are newly intubed, will receive UV light treatment to reduce SARS-CoV-2 viral load.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed positive test result for SARS-CoV-2
* Mechanically ventilated
* Endotracheal tube inner diameter of at least 7.5 mm

Exclusion Criteria:

* Unable to provide informed consent (or surrogate)
* Enrolled in a therapeutic clinical trial for same condition that does not allow recruitment in other trials
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Chaux, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rezaie A, Melmed GY, Leite G, Mathur R, Takakura W, Pedraza I, Lewis M, Murthy R, Chaux G, Pimentel M. Endotracheal Application of Ultraviolet A Light in Critically Ill Patients with Severe Acute Respiratory Syndrome Coronavirus 2: A First-in-Human Study. Adv Ther. 2021 Aug;38(8):4556-4568. doi: 10.1007/s12325-021-01830-7. Epub 2021 Jun 26. PMID 34173969
- See also: Peer-reviewed publication — https://pubmed.ncbi.nlm.nih.gov/34173969/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Endotracheal UV Light
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Endotracheal UV Light
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Negative Change in Viral Load
Description: Change of viral load in upper airway in patients admitted to hospital for COVID-19
Time Frame: 5 days
Measure: Mean (Full Range); unit: log10 copies/mL
Arm/Group | Endotracheal UV Light
Number analyzed (Participants) | 5
log10 copies/mL | 3.2 [1.20 to 6.77]

2. Secondary Outcome: Change in Bacterial Load
Description: Change of bacterial load in upper airway
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: Colony forming units/mL
Arm/Group | Endotracheal UV Light
Number analyzed (Participants) | 5
Colony forming units/mL | 102000 (594000)

3. Secondary Outcome: Ventilated Associated Pneumonia
Description: Percentage of patients developing ventilated pneumonia (VAP) within 30 days of treatment
Time Frame: 1 month
Population: One case of probable ventilator associated pneumonia with purulent endotracheal secretions and positive endotracheal culture for Pseudomonas aeruginosa.
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal UV Light
Number analyzed (Participants) | 5
Participants | 1

4. Secondary Outcome: Days to Extubation
Description: Number of days patient is intubated with endotracheal tube or tracheostomy
Time Frame: 1 month
Population: Mean days of intubation within the first 30 days of therapy. Deceased patient was not included.
Measure: Mean (Full Range); unit: days
Arm/Group | Endotracheal UV Light
Number analyzed (Participants) | 4
days | 20.75 [6 to 30]

5. Secondary Outcome: Days to Discharge
Description: Number of days patient is discharged from the hospital
Time Frame: 1 month
Population: Mean number days for the patients to be discharged from the hospital within the first 30 days. Deceased patient was not included.
Measure: Mean (Full Range); unit: days
Arm/Group | Endotracheal UV Light
Number analyzed (Participants) | 4
days | 27.25 [19 to 30]

6. Secondary Outcome: Change in C-reactive Protein
Description: Change in C-reactive protein from baseline to the end of the treatment
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Endotracheal UV Light
Number analyzed (Participants) | 5
mg/L | 95.00 (48.00)

7. Secondary Outcome: Change in the World Health Organization (WHO) Coronavirus Disease (COVID)-19 10-point Ordinal Severity Scale by 30 Days
Description: The World Health Organization (WHO) COVID-19 10-point ordinal severity scale:
  0 uninfected, No viral RNA detected
  1. Asymptomatic; viral RNA detected
  2. Ambulatory Mild disease: Symptomatic; independent
  3. Ambulatory Mild disease: Symptomatic; assistance needed
  4. Hospitalized: Moderate disease; no oxygen therapy
  5. Hospitalized: Moderate disease; oxygen by mask or nasal prongs
  6. Hospitalized: sever disease, Oxygen by non-invasive ventilation or high flow
  7. Hospitalized: severe disease, intubation and mechanical ventilation, pO2/FiO2>=150 or SpO2/FiO2>=200
  8. Hospitalized: severe disease, Mechanical ventilation pO2/FiO2<150(SpO2/FiO2 <200) or vasopressors
  9. Hospitalized: severe disease, Mechanical ventilation pO2/FiO2<150 and vasopressors, dialysis or extracorporeal membrane oxygenation
  10. Death
Time Frame: 1 month
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Endotracheal UV Light
Number analyzed (Participants) | 5
Scores on a scale | 3.6 [-1 to 7]

8. Secondary Outcome: Catheter Tip Assessment on the Last Day of Treatment
Description: Assessment of total bacterial load on the UV catheter tip on the last day of treatment
Time Frame: 5 days
Population: Catheter tips could not be retrieved in a sterile fashion due to infectious disease protocols in ICU. Therefore, data were not collected.
Arm/Group | Endotracheal UV Light
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 30 following enrollment.
Description: No treatment-emergent adverse events or need for treatment cessation was observed in the study. Oxygen saturations and hemodynamics during all treatment sessions remained stable. No subject experienced pneumothorax, subcutaneous emphysema, or ET tube dislodgment. All subjects survived except study subject 2, who was placed on comfort care following ICH due to ECMO-associated anticoagulation and died on ICU day 17. This complication was not related to study treatment.
Groups:
- Endotracheal UV Light: Mechanically ventilated patients who will receive UV Light therapy
  UV Light Treatment: UV light therapy administered while patient is mechanically ventilated
  No treatment-emergent adverse events or need for treatment cessation was observed in the study. Oxygen saturations and hemodynamics during all treatment sessions remained stable. None of the subjects experienced pneumothorax, subcutaneous emphysema, venous thromboembolism, or endotracheal tube (ETT) dislodgment.
Arm/Group | Endotracheal UV Light
All-Cause Mortality (participants affected / at risk) | 1/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT04572399/Prot_SAP_001.pdf